CLINICAL TRIAL: NCT01470846
Title: Epidural Analgesia vs. Morphine Patient-controlled Analgesia in Abdominal Surgery Under Laparotomy : a Medico-economic Study
Brief Title: Postoperative Analgesia in Abdominal Surgery: a Medico-economic Study
Acronym: PERIDIGE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patients eligible for the study
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I10030 PERIDIGE
Record Dates: First submitted 2011-11-08; First posted 2011-11-11 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Extended Ileal Resection Under Laparotomy; Total Proctocolectomy Under Laparotomy; Colectomy Left/Right/Total Under Laparotomy; Rectosigmoidal Resection Under Laparotomy; Anterior Resection of Rectum Under Laparotomy; Abdomino-perineal Amputation Under Laparotomy
Keywords: epidural analgesia; morphin analgesia; laparotomy
MeSH Terms: interventions — Analgesia, Epidural; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- APD (Experimental): patient with epidural analgesia
  Interventions: Procedure: epidural analgesia
- PCA (Active Comparator): Patient with morphine analgesia
  Interventions: Procedure: PCA

INTERVENTIONS:
Procedure: epidural analgesia — thoracic position (T8-T9 or T11-T12) depending on the site of surgery
  Arms: APD
Procedure: PCA — Morphine 2 mg / 10 min (no max dose) + droperidol 2.5 mg / 50 mL.
  Arms: PCA

SUMMARY:
Background : Epidural anaesthesia is associated in abdominal surgery with reduced pain and postoperative respiratory complications together with quicker recovery of bowel function. Currently, no studies have been able to prove its ability to reduce length of stay in intensive care and high-dependency units.

Purpose : The aim of this study is to demonstrate that epidural anaesthesia reduces length of stay in intensive care unit after abdominal surgery under laparotomy.

DETAILED DESCRIPTION:
There are currently two methods of analgesia in postoperative abdominal surgery : patient-controlled analgesia (PCA) with opioids and epidural analgesia.

No international recommendations regarding the use of either of these techniques have yet been written. Epidural analgesia is superior to intravenous morphine, including during mobilization and coughing. It also reduces respiratory complications and optimizes postoperative rehabilitation. Nevertheless, mortality is not improved with this technique. Few publications exist on the optimization of the duration of hospitalization in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Surgery scheduled under laparotomy
* Extended ileal resection
* Total proctocolectomy
* Colectomy left/right/total
* Rectosigmoidal resection
* Anterior resection of rectum
* Abdomino-perineal amputation
* Adult patient
* Written consent obtained
* Planned hospitalization in the intensive care unit
* Patient affiliated to social security

Exclusion Criteria:

* Patients inapt to give consent
* Emergency surgery
* Contraindication to epidural analgesia
* Contraindication to levobupivacaïne, morphine or sufentanil
* Dementia
* Participation in another research protocol
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Theoretical duration of hospitalization in intensive care unit. | 5 days
  The difference between the day of surgery and the day when discharge criteria for intensive care unit are met.

SECONDARY OUTCOMES:
Total duration of hospitalization. | 9 days
  The difference between the day of surgery and the day when the discharge criteria are met

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie NATHAN-DENIZOT, MD, Principal Investigator — Limoges UH
Locations (1):
- CHU de Limoges - Service d'anesthésie-réanimation, Limoges, France